CLINICAL TRIAL: NCT05541133
Title: Effect of Acute Exercise on Exosome Associated Biomarkers
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, K. Sreekumaran Nair, Principal Investigator, Mayo Clinic
Other Study IDs: 22-000001
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples collected before, during, and after acute exercise.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This research study is being done to understand the underlying mechanism by which exercise affects the body on the cellular level, in an acute aerobic endurance setting. This may help to better understand the overall benefits of endurance exercise.

ELIGIBILITY:
Inclusion Criteria:

* Ages: 18 to 45 years

Exclusion Criteria:

* BMI >32 kg/m2. Cardiovascular, metabolic (type 2 diabetes, fasting plasma glucose at or above 110 mg/dL and untreated hypo- or hyperthyroidism) or renal disease.
* Orthopedic problems that would keep them from being able to perform an exercise. - --
* Medications that are known to affect mitochondrial function: Corticosteroids, opiates, benzodiazepines, tricyclic antidepressants, beta-blockers, sulfonylureas, insulin, anticoagulants, barbiturates, insulin sensitizers, fibrates (PPAR gamma agonist).
* Smoking.
* Pregnancy.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Generally healthy individuals around the Rochester MN area.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2022-07-09 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
List of biomarkers | Baseline
  Exosome proteomes and MiRNA from blood samples

CONTACTS AND LOCATIONS:
Overall Officials: K. Sreekumaran Nair, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials